CLINICAL TRIAL: NCT01760070
Title: Comparison of O-type Hybrid Knife and IT Knife in Endoscopic Submucosal Dissection for Upper Gastrointestinal Neoplasms: a Prospective Randomized Controlled Trial
Brief Title: Comparison of O-type Hybrid Knife and IT Knife in ESD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhiguo Liu, Associate Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XIJINGHDD-20121227-01
Record Dates: First submitted 2012-12-28; First posted 2013-01-03 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Esophageal Cancer; Esophageal Dysplasia; Stomach Cancer; Stomach Dysplasia
Keywords: cancer; endoscopy; endoscopic submucosal dissection
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hybrid knife (Experimental): O-type Hybrid knife is used the whole ESD process except for minimum use of dual knife in border marking and initial mucosal cutting.
  Interventions: Device: Hybrid knife
- IT knife (Active Comparator): IT knife is used the whole ESD process except for minimum use of dual knife in border marking and initial mucosal cutting.
  Interventions: Device: IT knife

INTERVENTIONS:
Device: Hybrid knife — Use Hybrid knife in ESD procedure
  Arms: Hybrid knife
Device: IT knife — Use IT knife in ESD procedure.
  Arms: IT knife

SUMMARY:
By combining injection and dissection capability together, O-type Hybrid knife could possibly shorten the endoscopic submucosal dissection procedure for upper gastrointestinal neoplasms.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) has been accepted as an minimal invasive alternative to surgery for localized early upper gastrointestinal neoplasms recently. However, the procedure remains to be technically challenging and time consuming. Many modified methods or newly developed devices were developed to simplify the procedure. A new insulated tip dissecting knife (O-type Hybrid knife) has been recently developed with both injection and lateral cutting capability. The aim of this study was to investigate whether ESD procedure could be shortened with this new device.

ELIGIBILITY:
Inclusion Criteria:

* Gastric or esophageal adenoma or early cancer which is eligible for conventional ESD indications
* The patients who agreed informed consent

Exclusion Criteria:

* Recent drug history of anticoagulant or antiplatelet agent within 7 days
* Recurrent gastric or esophageal adenoma or early cancer
* Pregnant or breast feeding patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Procedure time for ESD | up to 1 day
  The time to finish the whole ESD procedure.

SECONDARY OUTCOMES:
Submucosal dissection time | up to 1 day
  The time for submucosal dissection of ESD
Perforation rate | up to 7 day
  The perforation rate of ESD during and after procedure.
Bleeding Rate | up to 7 days
  The bleeding rate of ESD during and after procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Liu, Principal Investigator — Xijing Hospital of Digestive Diseases
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Lingenfelder T, Fischer K, Sold MG, Post S, Enderle MD, Kaehler GF. Combination of water-jet dissection and needle-knife as a hybrid knife simplifies endoscopic submucosal dissection. Surg Endosc. 2009 Jul;23(7):1531-5. doi: 10.1007/s00464-009-0433-3. Epub 2009 Apr 3. PMID 19343433
- [Background] Fukami N, Ryu CB, Said S, Weber Z, Chen YK. Prospective, randomized study of conventional versus HybridKnife endoscopic submucosal dissection methods for the esophagus: an animal study. Gastrointest Endosc. 2011 Jun;73(6):1246-53. doi: 10.1016/j.gie.2010.12.004. Epub 2011 Feb 12. PMID 21316668